CLINICAL TRIAL: NCT00429689
Title: Hormonal Levels in Men With Major Depressive Disorder
Status: Withdrawn | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Amiaz Revital, MD, Sheba Medical Center
Other Study IDs: SHEBA-06-4480-RA-CTIL
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Depression
Keywords: Male, MDD, Testosterone, DHEA-S,Cortisol; Male; 18-65; Major Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Saliva sample

SUMMARY:
Subjects will be 1000 men meeting the following inclusion criteria: 1) male, age 18-65 years; 2) meeting DSM-IV criteria for major depressive disorder within the past one year, with a HAM-D score >12.

Subjects will be excluded if they exhibit 1) a substance abuse or dependence disorder within the past year; 2) current psychotic symptoms; or 3) a history of bipolar disorder.

Procedure

After informed consent, eligible patients will have blood drawn for serum hormone levels; cortisol, DHEA-S and testosterone or they will provide a salivary sample for measurement of hormone levels.

We will also test hormone level form 1000 healthy males (from blood or saliva) at the same age for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Major Depression Disorder
* 18-65

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men diagnosed with Major depression disorder
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Seidman,, MD, Study Director — West End Medical Associates; Revital Amiaz, MD, Principal Investigator — Sheba Medical Center